CLINICAL TRIAL: NCT00335426
Title: Influence of Spinal Manipulative Therapy Upon Stroop Task Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Logan College of Chiropractic (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RD0601060018
Record Dates: First submitted 2006-06-07; First posted 2006-06-09 (Estimated); Last update posted 2009-09-01 (Estimated); Status verified 2009-08

CONDITIONS: Motor Response Time

INTERVENTIONS:
Procedure: Spinal manipulative therapy

SUMMARY:
The purpose of this study is to determine if spinal manipulative therapy can affect cognitive processing as determined by performance on a Stroop task. It is specifically hypothesized that number of errors and response times will decrease as a result of spinal manipulative therapy.

ELIGIBILITY:
Inclusion Criteria:

Normal healthy

Exclusion Criteria:

No spinal manipulation one week proceeding trial No stimulants or depressants

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2006-06; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristan J Giggey, DC, Principal Investigator — Logan College of Chiropractic
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States